CLINICAL TRIAL: NCT00515723
Title: Glucose and Lipid Metabolism on Antipsychotic Medication
Acronym: Glulipid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH063985-04 (NIH); R01MH063985-04 (NIH)
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Type 2 Diabetes Mellitus; Hyperglycemia
Keywords: control; risperidone; olanzapine; quetiapine; ziprasidone
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Diabetes Mellitus, Type 2; Hyperglycemia | interventions — Risperidone; Olanzapine; Quetiapine Fumarate; ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Olanzapine (Active Comparator): Participants in this group were randomized to flexibly-dosed treatment with olanzapine.
  Interventions: Drug: olanzapine
- Risperidone (Active Comparator): Participants in this group were randomized to flexibly-dosed treatment with risperidone.
  Interventions: Drug: risperidone
- Quetiapine (Active Comparator): Participants in this group were randomized to flexibly-dosed treatment with quetiapine.
  Interventions: Drug: quetiapine
- Ziprasidone (Active Comparator): Participants in this group were randomized to flexibly-dosed treatment with ziprasidone.
  Interventions: Drug: ziprasidone

INTERVENTIONS:
Drug: risperidone — randomized to 12 week trial of risperidone.
  Other Names: Risperdal
  Arms: Risperidone
Drug: olanzapine — randomized to 12 week trial of olanzapine.
  Other Names: Zyprexa
  Arms: Olanzapine
Drug: quetiapine — randomized to 12 week trial of quetiapine.
  Other Names: Seroquel
  Arms: Quetiapine
Drug: ziprasidone — randomized to 12 week trial of ziprasidone.
  Other Names: Geodon
  Arms: Ziprasidone

SUMMARY:
This project aims to a) evaluate the effects of selected antipsychotic medications on insulin action in skeletal muscle (glucose disposal), liver (glucose production) and adipose tissue (whole-body lipolysis), b) evaluate the effects of selected antipsychotic medications on abdominal adipose tissue mass, total body fat and total fat-free mass, and c) explore the longitudinal effects of treatment with selected antipsychotics on glucose tolerance, lipid profiles, abdominal adipose tissue mass, total body fat and total fat-free mass. These hypotheses will be evaluated by measuring 1) whole-body glucose and lipid kinetics with the use of "gold-standard" stable isotope tracer methodology, 2) body composition using dual energy x-ray absorptiometry and magnetic resonance imaging, and 3) longitudinal changes in glucose tolerance and lipid profiles. The aims will be addressed in non-diabetic schizophrenia patients chronically treated with risperidone, olanzapine, clozapine, quetiapine, ziprasidone, or haloperidol, and untreated healthy controls. Re-evaluations will also be performed in patients who are randomized to switch from their current antipsychotic (from the above groups) to risperidone, olanzapine, quetiapine, or ziprasidone for 6 months. Relevant data is critically needed to target basic research, identify long-term cardiovascular consequences, and plan therapeutic interventions.

DETAILED DESCRIPTION:
Hyperglycemia and type 2 diabetes mellitus are more common in schizophrenia than in the general population. Type 2 diabetes mellitus is characterized by disturbances in insulin action on skeletal muscle, liver and adipose tissue. Diabetes causes increased morbidity and mortality due to acute (e.g., diabetic ketoacidosis) and long-term (e.g., cardiovascular disease) complications. The combination of hyperglycemia, dyslipidemia and abdominal adiposity is even more strongly associated with increased cardiovascular morbidity and mortality. The association of type 2 diabetes and hyperglycemia with schizophrenia was first noted prior to the introduction of antipsychotic medications, suggesting that these patients may be at increased risk. Since then, however, additional glucoregulatory abnormalities (e.g., new onset diabetes), dyslipidemia, and increased weight and adiposity have all been associated with antipsychotic medications. Concern about antipsychotic effects on glucose, lipids and adiposity has increased recently, focusing on the widely-used newer medications, clozapine and olanzapine. Increased abdominal adiposity can secondarily decrease insulin sensitivity and antipsychotics can increase adiposity. However, medication effects on glucose control and insulin action may also occur independent of differences in adiposity. This project aims to a) evaluate the effects of selected antipsychotic medications on insulin action in skeletal muscle (glucose disposal), liver (glucose production) and adipose tissue (whole-body lipolysis), b) evaluate the effects of selected antipsychotic medications on abdominal adipose tissue mass, total body fat and total fat-free mass, and c) explore the longitudinal effects of treatment with selected antipsychotics on glucose tolerance, lipid profiles, abdominal adipose tissue mass, total body fat and total fat-free mass. These hypotheses will be evaluated by measuring 1) whole-body glucose and lipid kinetics with the use of "gold-standard" stable isotope tracer methodology, 2) body composition using dual energy x-ray absorptiometry and magnetic resonance imaging, and 3) longitudinal changes in glucose tolerance and lipid profiles. The aims will be addressed in non-diabetic schizophrenia patients chronically treated with risperidone, olanzapine, clozapine, quetiapine, ziprasidone, or haloperidol, and untreated healthy controls. Re-evaluations will also be performed in patients who are randomized to switch from their current antipsychotic (from the above groups) to risperidone, olanzapine, quetiapine, or ziprasidone for 6 months. Relevant data is critically needed to target basic research, identify long-term cardiovascular consequences, and plan therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years
* Patients: otherwise healthy and meets DSM-IV criteria for schizophrenia or schizoaffective disorder, any type, treated with haloperidol, olanzapine, clozapine, quetiapine, ziprasidone, aripiprazole, or risperidone for at least 3 months
* Controls: healthy
* Able to give informed consent
* No antipsychotic medication changes for 3 months, and no other medication changes for 2 weeks prior to Baseline Evaluations.

Exclusion Criteria:

* Axis I psychiatric disorder criteria met in self except for substance use disorders as below
* Patients and controls: meets DSM-IV criteria for the diagnoses of substance abuse within the past 3 months
* Involuntary legal status (as per Missouri law)
* The presence of any serious medical disorder that may confound the assessment of relevant biologic measures or diagnosis, including: significant organ system dysfunction, metabolic diseases, type 1 diabetes mellitus, symptomatic type 2 diabetes mellitus (see below), pregnancy, endocrine disease, coagulopathy, clinically significant anemia, that would preclude blood sampling (as determined by the PI) or acute infection;
* Patients taking more than one atypical antipsychotic medication;
* Subjects taking certain prescription medications (as determined by PI on a case by case basis).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2001-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W Newcomer, MD, Principal Investigator — Washington Univerisity School of Medicine and Florida Atlantic University
Locations (2):
- United States (2):
  - Washington Univeristy School of Medicine, St Louis, Missouri
  - Washington University School of Medicine, Psychiatry Dept., St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from wide range of sites in the St. Louis community. Some advertising with flyers was used however the majority of the recruitment was done using community outreach,doctor-to-doctor or self-referrals, and referrals from board and care and community support programs. All recruitment materials were approved by the IRB.
Pre-assignment Details: Participants were enrolled in the study once they signed consent. After enrollment, participants were brought in for a screening visit consisting of a diagnostic interview, screening labs, a review of records and a discussion with their primary psychiatrist. If the patient met all inclusion criteria after screening, study visits were scheduled.
Period: Overall Study
Arm/Group | Olanzapine | Risperidone | Quetiapine | Ziprasidone
Started | 25 | 22 | 22 | 27
Completed | 20 | 21 | 21 | 21
Not Completed | 5 | 1 | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Olanzapine: Participants with schizophrenia were randomized to olanzapine.
- Risperidone: Patients with schizophrenia were randomized to risperidone.
- Quetiapine: Participants with schizophrenia were randomized to quetiapine.
- Ziprasidone: Participants with schizophrenia were randomized to ziprasidone.
- Total: Total of all reporting groups
Arm/Group | Olanzapine | Risperidone | Quetiapine | Ziprasidone | Total
Number analyzed (Participants) | 25 | 22 | 22 | 27 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (11.2) | 39.2 (11.1) | 36.4 (8.6) | 38.3 (10.2) | 37.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 9 | 11 | 31
  Male | 18 | 18 | 13 | 16 | 65
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 7 | 4 | 11 | 30
  Non-White | 17 | 15 | 17 | 16 | 65
  Unknown | 0 | 0 | 1 | 0 | 1
Body Weight [Mean (Standard Deviation); unit: kilograms] | 98.75 (21.04) | 93.88 (19.19) | 92.95 (18.67) | 94.68 (15.90) | 95.16 (18.56)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per squared meters] | 32.27 (7.38) | 31.04 (6.50) | 31.76 (6.63) | 32.27 (5.56) | 31.87 (6.45)
Waist Circumference [Mean (Standard Deviation); unit: centimeters] | 108.44 (16.74) | 102.87 (16.66) | 104.10 (15.45) | 108.50 (15.18) | 106.19 (15.95)
DEXA Total Fat [Mean (Standard Deviation); unit: kilograms] — Population: 3 participants were missing a baseline DEXA scan.
  kilograms
    number analyzed (Participants) | 25 | 20 | 21 | 27 | 93
    (all) | 32.24 (13.49) | 24.95 (10.07) | 28.69 (11.63) | 31.60 (11.22) | 29.68 (11.89)
Whole Body Sensitivity [Mean (Standard Deviation); unit: mg/kg/min] — Population: Two participants were missing data due to bad veins.
  mg/kg/min
    number analyzed (Participants) | 24 | 21 | 22 | 27 | 94
    (all) | 4.39 (2.16) | 5.53 (3.32) | 5.10 (2.93) | 4.33 (2.01) | 4.79 (2.62)

OUTCOME MEASURES:

1. Primary Outcome: DEXA Total Fat
Description: This study hypothesized that antipsychotic treatment would increase total body fat, as measured by whole body dual energy x-ray absorptiometry (DEXA), with larger adverse effects for olanzapine.
Time Frame: The relevant time points include baseline, week 6 and week 12.
Population: Modified Intent to Treat (ITT) sample with week 0, week 6 and week 12 data. Two Quetiapine participants were excluded from analyses due to failure to adhere to the protocol.
Measure: Mean (Standard Error); unit: kilograms of body fat
Groups:
- Total: This arm consists of all treatments pooled together.
Arm/Group | Olanzapine | Risperidone | Quetiapine | Ziprasidone | Total
Number analyzed (Participants) | 25 | 22 | 20 | 27 | 94
kilograms of body fat
  Baseline | 32.24 (2.48) | 27.66 (2.64) | 28.83 (2.77) | 31.60 (2.38) | 30.25 (1.27)
  6 Weeks | 34.38 (2.48) | 28.29 (2.64) | 29.60 (2.77) | 31.18 (2.39) | 31.05 (1.27)
  12 Weeks | 35.45 (2.49) | 29.23 (2.64) | 30.10 (2.77) | 30.66 (2.40) | 31.52 (1.28)
Statistical Analysis 1: Comparison: Total; Primary analysis for change in DEXA total fat used a likelihood-based mixed-effects model using time (0, 6, and 12 weeks) as the independent variable, with Toeplitz covariance structure specified, based on Akaike Information Criterion-Corrected (AIC-C). The null hypothesis was that there was no difference in the outcome over time (main effect of time); Test type: Superiority; p = 0.002, Mixed Models Analysis — The a priori threshold for statistical significance in this planned primary test was p<0.05
Statistical Analysis 2: Comparison: Olanzapine vs Risperidone vs Quetiapine vs Ziprasidone; Primary analysis for change in DEXA total fat used a likelihood-based mixed-effects model using time (0, 6, and 12 weeks) and treatment group as independent variables, with Toeplitz covariance structure specified, based on Akaike Information Criterion-Corrected (AIC-C). The null hypothesis was that there were no differences between groups in the change over time (time by treatment condition); Test type: Superiority; p = 0.002, Mixed Models Analysis — The a priori threshold for statistical significance in this planned primary test was p<0.05

2. Primary Outcome: Clamp Derived Insulin Sensitivity (mg/kg/Min)
Description: This study hypothesized that antipsychotic treatment would decrease insulin sensitivity, with larger adverse effects for olanzapine. Insulin sensitivity describes how sensitive the body is to the effects of insulin.
Time Frame: The relevant time points include baseline and week 12.
Population: Modified Intent to Treat (ITT) sample with Week 0 and Week 12 data. Two Quetiapine participants were excluded from analyses due to failure to adhere to the protocol.
Measure: Mean (Standard Error); unit: mg/kg/min
Arm/Group | Olanzapine | Risperidone | Quetiapine | Ziprasidone | Total
Number analyzed (Participants) | 25 | 22 | 20 | 27 | 94
mg/kg/min
  Baseline | 4.39 (0.53) | 5.53 (0.57) | 5.28 (0.58) | 4.33 (0.50) | 4.82 (0.27)
  Week 12 | 3.62 (0.49) | 5.01 (0.51) | 5.08 (0.53) | 4.45 (0.47) | 4.50 (0.25)
Statistical Analysis 1: Comparison: Total; Primary analysis for change in insulin sensitivity used a likelihood-based mixed-effects model using time (0 and 12 weeks) as the independent variable, with an unstructured covariance structure specified, based on the Akaike Information Criterion-Corrected (AIC-C). The null hypothesis was that there was no difference in the outcome over time (main effect of time); Test type: Superiority; p = 0.05, Mixed Models Analysis — The a priori threshold for statistical significance in this planned primary test was p<0.05
Statistical Analysis 2: Comparison: Olanzapine vs Risperidone vs Quetiapine vs Ziprasidone; Primary analysis for change in insulin sensitivity used a likelihood-based mixed-effects model using time (0 and 12 weeks) and treatment group as the independent variables, with an unstructured covariance structure specified, based on the Akaike Information Criterion-Corrected (AIC-C). The null hypothesis was that there were no differences between groups in the change over time (time by treatment condition); Test type: Superiority; p = 0.22, Mixed Models Analysis — The a priori threshold for statistical significance in this planned primary test was p<0.05

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study's primary time points, baseline and week 12. However, only adverse events at week 12 are provided as these are potentially related to the treatments. As a result, the sample sizes differ from the sample sizes found in the Participant Flow section as not everyone made it to week 12.
Arm/Group | Olanzapine | Risperidone | Quetiapine | Ziprasidone
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21 | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21 | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 13/19 | 8/21 | 9/20 | 11/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olanzapine (N=19) | Risperidone (N=21) | Quetiapine (N=20) | Ziprasidone (N=21)
Drowsiness/Somnolence (Psychiatric disorders) | 9 | 3 | 5 | 6
Tiredness/Fatigue (Psychiatric disorders) | 8 | 4 | 4 | 4
Hunger (Psychiatric disorders) | 5 | 3 | 3 | 2
Anxiety (Psychiatric disorders) | 1 | 2 | 2 | 2
Restlessness (Psychiatric disorders) | 1 | 1 | 1 | 3
Headache (Psychiatric disorders) | 1 | 1 | 3 | 0
Difficulty Concentrating (Psychiatric disorders) | 0 | 0 | 0 | 3
Tremor (Psychiatric disorders) | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No